CLINICAL TRIAL: NCT02459457
Title: A Comparison of Paclitaxel in Combination With Cisplatin(TP), Carboplatin(TC) or Fluorouracil(TF) Concurrent With Radiotherapy for Patients With Local Advanced Esophageal Squamous Cell Carcinoma: A Three-Arm Randomized Phase III Trial
Brief Title: A Comparison of Paclitaxel-based Three Regimens Concurrent With Radiotherapy for Patients With Local Advanced Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Huadong Hospital (Other); Wuxi No. 4 People's Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Jiangxi Provincial Cancer Hospital (Other); Shanxi Province Cancer Hospital (Other); Gansu Cancer Hospital (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai 2
Record Dates: First submitted 2015-05-23; First posted 2015-06-02 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Stage III Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; concurrent chemoradiotherapy; paclitaxel; cisplatin; carboplatin; fluorouracil
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — TP protocol; Paclitaxel; Fluorouracil; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Paclitaxel and Cisplatin (TP) (Active Comparator): Patients receive TP concurrent with radiotherapy (1.8Gy/d, d1-5/week, 34Fx) Paclitaxel: 175mg/m2/d, ivgtt over 3 hours, d1; Cisplatin: 25mg/m2/d, ivgtt, d1-3, q4w*4
  Interventions: Drug: Paclitaxel and Cisplatin; Radiation: Radiotherapy
- Paclitaxel and Fluorouracil (TF) (Active Comparator): Patients receive TF concurrent with radiotherapy(1.8Gy/d, d1-5/week, 34Fx) Concurrent: paclitaxel 50mg/m2/d, ivgtt over 3 hours, d1; 5-FU 300mg/m2, civ 96h, d1-4, qw*6; Adjuvant: paclitaxel 175 mg/m2/d, ivgtt over 3 hours, d1; 5-FU 1800mg/m2, civ 72h, d1-3, q4w*2
  Interventions: Drug: Paclitaxel and Fluorouracil; Radiation: Radiotherapy
- Paclitaxel and Carboplatin（TC） (Active Comparator): Patients receive TC concurrent with radiotherapy(1.8Gy/d, d1-5/week, 34Fx) Concurrent: paclitaxel 50mg/m2/d, ivgtt over 3 hours, d1; carboplatin AUC=2, ivgtt, d1, qw*6; Adjuvant: paclitaxel 175 mg/m2/d, ivgtt over 3 hours, d1; carboplatin AUC=5, ivgtt, d1, q4w*2
  Interventions: Drug: Paclitaxel and Carboplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Paclitaxel and Cisplatin — patients get Paclitaxel and Cisplatin according to protocol
  Other Names: TP
  Arms: Paclitaxel and Cisplatin (TP)
Drug: Paclitaxel and Fluorouracil — patients get Paclitaxel and Fluorouracil according to protocol
  Other Names: TF
  Arms: Paclitaxel and Fluorouracil (TF)
Drug: Paclitaxel and Carboplatin — patients get Paclitaxel and Carboplatin according to protocol
  Other Names: TC
  Arms: Paclitaxel and Carboplatin（TC）
Radiation: Radiotherapy — 1.8Gy/d, d1-5/week, 34Fx

SUMMARY:
The purpose of this study is to determined the best scheme in paclitaxel and cisplatin，paclitaxel and fluorouracil，paclitaxel and carboplatin concurrent with radiotherapy for patients with local advanced esophageal Squamous Cell Carcinoma.

ELIGIBILITY:
Inclusion criteria

To be eligible for this study, patient must fulfill all of the following criteria:

1. Histologically confirmed esophageal squamous cell carcinoma
2. Clinical stages II, III or IVa based on the 6th UICC-TNM classification
3. No prior treatment of chemotherapy, radiotherapy or surgery against esophageal cancer, except for non-curative resection by EMR/ESD.
4. Aged 18-75 years
5. Adequate organ functions

   1. White blood cell (WBC) ≥3×109⁄L
   2. Absolute neutrophil counts (ANC) ≥1.5×109⁄L
   3. Hemoglobin (Hb) ≥10g⁄dl
   4. Platelet (Plt) ≥100×109⁄L
   5. Total bilirubin <1.5 upper limit of normal (ULN)
   6. Aspartate transaminase (AST) ≤2.5 ULN
   7. Alanine aminotransferase (ALT) ≤2.5 ULN
   8. Creatinine ≤1.5 ULN
6. ECOG PS of 0-2
7. Life expectancy ≥3 months
8. Written informed consent

Exclusion criteria Patients fulfilling any of the following criteria are ineligible for this study.

1. Esophageal perforation or hematemesis
2. Synchronous or metachronous malignancies (except for cutaneous (non-melanomas) carcinoma, thyroid papillary carcinoma, phase I seminoma or cervical carcinoma in situ curatively treated and disease free for a minimum of 3 months)
3. Received thoracic, abdominal or craniocerebral surgery within 30 days
4. Enrolled in other clinical trials within 30 days
5. Unstable angina and/or congestive heart failure requiring hospitalization within 6 months
6. Severe psychiatric disease
7. Pregnancy, lactation or unwillingness to adopt contraception
8. Drug addiction
9. Acquired immune deficiency syndrome (AIDS) based upon current CDC definition
10. Patients with hearing impairment or sensory-motor neuropathy of WHO grade > 1
11. History of radiotherapy in the planning area
12. Other ineligible conditions according to researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
overall survival | 3 years

SECONDARY OUTCOMES:
progression free survival | 1year, 2 years, 3 years
adverse event | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kuaile Zhao, MD, Study Chair — +86 18017312534
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ai D, Ye J, Wei S, Li Y, Luo H, Cao J, Zhu Z, Zhao W, Lin Q, Yang H, Zheng X, Zhou J, Huang G, Li L, Li J, Zhang Z, Zhou G, Gu D, Du M, Mo M, Jia H, Zhang Z, Zhao K. Comparison of 3 Paclitaxel-Based Chemoradiotherapy Regimens for Patients With Locally Advanced Esophageal Squamous Cell Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e220120. doi: 10.1001/jamanetworkopen.2022.0120. PMID 35188552
- [Derived] Ai D, Chen Y, Liu Q, Zhang J, Deng J, Zhu H, Ren W, Zheng X, Li Y, Wei S, Ye J, Zhou J, Lin Q, Luo H, Cao J, Li J, Huang G, Wu K, Fan M, Yang H, Zhu Z, Zhao W, Li L, Fan J, Badakhshi H, Zhao K. Comparison of paclitaxel in combination with cisplatin (TP), carboplatin (TC) or fluorouracil (TF) concurrent with radiotherapy for patients with local advanced oesophageal squamous cell carcinoma: a three-arm phase III randomized trial (ESO-Shanghai 2). BMJ Open. 2018 Oct 21;8(10):e020785. doi: 10.1136/bmjopen-2017-020785. PMID 30344165